CLINICAL TRIAL: NCT05696613
Title: A Phase 3 Superiority Study Comparing the Safety and Efficacy of SNP-ACTH (1-39) Gel Compared to Rituximab and FDA Approved Biosimilars in Adults With Primary Membranous Nephropathy (PMN) in a Two-Phase Adaptive Trial Design
Brief Title: A Study of SNP-ACTH (1-39) Gel in Patients With Primary Membranous Nephropathy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cerium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTH-PMN-301
Record Dates: First submitted 2022-12-29; First posted 2023-01-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Primary Membranous Nephropathy
Keywords: Kidney disease; Rituximab; Nephritis; Melanocortin; Hormones; Glucocorticoids; Glomerular Disease; ACTH; PMN
MeSH Terms: conditions — Kidney Diseases; Nephritis | interventions — Gels; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 3a Cohort 1 (Experimental): 3 mg SNP-ACTH Gel sc injection 3 times per week
  Interventions: Drug: SNP-ACTH (1-39) Gel
- Phase 3a Cohort 2 (Experimental): 5 mg SNP-ACTH Gel sc injection 3 times per week
  Interventions: Drug: SNP-ACTH (1-39) Gel
- Phase 3b Cohort 1 (Experimental): Dose level to be confirmed once Phase 3a part is completed
  Interventions: Drug: SNP-ACTH (1-39) Gel
- Phase 3b Cohort 2 (Active Comparator): Rituximab arm: Patients randomized to the rituximab arm will receive 1 g IV infusion on T0 (after baseline measures are collected) and day 15. A second course of rituximab 1g IV infusion will be administered 6 months after the first rituximab infusion and an additional 1 g IV infusion 14 days following the first 6-month infusion.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: SNP-ACTH (1-39) Gel — Subjects will be randomly assigned in 1:1 treatment allocation ratio to receive the test and reference product.
  Arms: Phase 3a Cohort 1; Phase 3a Cohort 2; Phase 3b Cohort 1
Drug: Rituximab — Subjects will be randomly assigned in 1:1 treatment allocation ratio to receive the test and reference product.
  Other Names: Rituxan or other biosimilars
  Arms: Phase 3b Cohort 2

SUMMARY:
The goal of the Phase 3a part of this clinical trial is to determine the optimal dose that will be used in the Phase 3b part of this clinical trial. The goal of the Phase 3b part is to assess the efficacy of SNP-ACTH (1-39) Gel relative to rituximab in patients with primary membranous nephropathy (PMN) at month 24.

DETAILED DESCRIPTION:
This head-to-head, open-label, 2-phase superiority trial compares SNP-ACTH (1-39) Gel to rituximab in the treatment of PMN that commences with an adaptive trial design for dose finding. The trial will be divided into 2 parts: Phase 3a and Phase 3b.

Dose finding Phase 3a part of the study will enroll a total of 16 patients randomized to 2 different dose levels of SNP-ACTH (1-39) Gel treatment for 12 months. Dose levels will be:

* 8 patients at 3mg SNP-ACTH Gel subcutaneous (sc) injection 3 times per week;
* 8 patients at 5mg SNP-ACTH Gel sc injection 3 times per week

Data from the Phase 3a part of the study will be assessed at regular intervals (at months 2, 3, 4, 5, 6, 9, 12) and will inform the dose selection for the Phase 3b. The optimal dose will be determined based on a risk/benefit assessment from data obtained from the Phase 3a part of the study, with the earliest assessment being conducted after all patients have completed at least 2 months of therapy.

The Phase 3b part of the study will enroll 132 patients randomized 1:1 to either 12 months of 1g Rituximab therapy (2 treatment cycles at month 1 and month 6) or 12 months of SNP-ACTH (1-39) Gel treatment at the dose level determined in the Phase 3a.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven membranous glomerulonephritis or a diagnosis of MN in patients with Nephrotic Syndrome and a positive anti PLA2R antibody test.
* Patients classified to be at a High Risk for progressive loss of kidney function, as defined by Kidney Disease Improving Global Outcomes (KDIGO) 2021-Glomerular Diseases Guideline.
* eGFR by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula ≥40 mL/min/1.73 m^2
* Patients who have had CR or PR in response to immunosuppressive therapy, but then relapsed can participate in the study if it has been more than 3 months since their last dose of high dose glucocorticoids, calcineurin inhibitors or mycophenolate mofetil
* Patients who have had CR or PR in response to IS therapy, but then relapsed can participate in the study if it has been more than 6 months since their last dose of chlorambucil or cyclophosphamide
* Patients who have had CR or PR in response to immunosuppressive therapy, but then relapsed can participate in the study if it has been more than 12 months since their last dose of rituximab.
* Life expectancy > 24 months.
* Other inclusion criteria may apply.

Exclusion Criteria:

* Secondary membranous nephropathy as defined by history, physical exam, kidney biopsy results or serologies.
* Patients who have had a ≥ 50% reduction in serum titers of PLA2R auto-antibody within 1 year before screening.
* Type 1 or 2 diabetes mellitus
* Patients who must be initiated on drugs likely to affect renal function if not properly dosed.
* Surgery within 1 month of study entry
* History of sensitivity to proteins of porcine origin.
* Other exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in urinary protein (Phase 3a) | Change from baseline, months 1, 2, 3, 4, 5, 6, 9, and 12
Change in Anti-phospholipase A2 receptor (PLA2R) auto-antibody levels (Phase 3a) | Change from baseline, months 1, 2, 3, 4, 6, and 12
Complete response of PMN (Phase 3b) | 24 months
  Reduction of proteinuria to ≤0.3 g/24 hours as measured by urine protein/creatinine ratio obtained from a 24-hour urine collection with stable renal function defined as a <15% decline in eGFR at the time of endpoint assessment

SECONDARY OUTCOMES:
Relapse rate at month 12 and month 24. | 12 and 24 months
Anti-PLA2R (or Anti-THSD7A) auto-antibody levels. | 12 and 24 months
Estimated glomerular filtration rate (eGFR) with proteinuria levels. | 12 and 24 months
Adverse events | 24 months
Incidence of ADAs | 24 months
Number of patients who achieved a complete remission (CR) or partial remission (PR) at month 12. | 12 months
Number of patients who achieved a Immunological Response (IR) at month 12. | 12 months
Assessment of time to achieving CR, PR, IR. | 24 months
Assessment of time to relapse for patients who achieved CR, PR, IR. | 12 and 24 months
Duration of time between initial achievement of CR to latest date of observed remission. | 24 months

CONTACTS AND LOCATIONS:
Locations (31):
- United States (19):
  - Academic Medical Research Institute, Los Angeles, California
  - North America Research Institute, San Dimas, California
  - Valiance Clinical Research, Tarzana, California
  - RecioMed Clinical Research Network, Inc., Boynton Beach, Florida
  - South Florida Nephrology Research, Coral Springs, Florida
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Reliant Medical Research, LLC, Miami, Florida
  - Vista Health Research, LLC, Miami, Florida
  - Genesis Clinical Research, Tampa, Florida
  - Fides Clinical Research, Atlanta, Georgia
  - Costal Medical Research, Brunswick, Georgia
  - Insight Hospital and Medical Center Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Center for Advanced Kidney Research, PLC, Saint Clair Shores, Michigan
  - NYU Langone Health, New York, New York
  - Prolato Clinical Research Center, Houston, Texas
  - P&I Clinical Research LLC, Lufkin, Texas
  - University of Virginia, Charlottesville, Virginia
  - Nephrology Associates of Northern Virginia, Fairfax, Virginia
- Regional Kidney Wellness Centre, Brampton, Ontario, Canada
- India (11):
  - Vedanta Hospitals, Guntur, Andhra Pradesh
  - Vijaya Super Speciality Hospital, Nellore, Andhra Pradesh
  - AIIMS, Raipur, Chhattisgarh
  - Muljibhai Patel Urological Hospital, Nadiād, Gujarat
  - KLE Hospital, Belagavi, Karnataka
  - Saraswati Kidney Care Center, Nagpur, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - PGIMER, Chandigarh, Punjab
  - SMS Medical College and Hospital, Jaipur, Rajasthan
  - Apex Hospitals, Jaipur, Rajasthan
  - Galaxy Hospital, Varanasi, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No